CLINICAL TRIAL: NCT02467400
Title: Dose Response and Receptor Selectivity of Beta-blocker Effects on Bone Metabolism
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Sundeep Khosla, M.D., Professor of Medicine and Physiology, College of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 14-004305
Record Dates: First submitted 2015-06-04; First posted 2015-06-10 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Osteoporosis, Age-Related
Keywords: bone formation
MeSH Terms: conditions — Osteoporosis | interventions — Atenolol; Nebivolol; Propranolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- placebo (Placebo Comparator): Sugar pill 2/day for 20 weeks; The once daily groups will receive a placebo as the second dose
  Interventions: Drug: placebo
- Atenolol (Active Comparator): Atenolol 50 mg 1/day for 20 weeks
  Interventions: Drug: Atenolol
- Nebivolol (Active Comparator): Nebivolol 5 mg/day for 20 weeks
  Interventions: Drug: Nebivolol
- Propranolol 40 mg (Active Comparator): Propranolol 20 mg bid for 20 weeks
  Interventions: Drug: Propranolol
- Propranolol 80 mg (Active Comparator): Propranolol 40 mg bid for 20 weeks
  Interventions: Drug: Propranolol

INTERVENTIONS:
Drug: Atenolol — beta blocker
  Arms: Atenolol
Drug: Nebivolol — beta blocker
  Arms: Nebivolol
Drug: Propranolol — beta blocker
  Arms: Propranolol 40 mg; Propranolol 80 mg
Drug: placebo — placebo
  Arms: placebo

SUMMARY:
This study is designed to answer the question as to whether the sympathetic nervous system is an important determinant of bone metabolism in humans.

DETAILED DESCRIPTION:
In postmenopausal women, who have increased sympathetic outflow, to test the hypothesis that treatment with low doses of a non-selective β-blocker (propranolol) will increase serum markers of bone formation and reduce markers of bone resorption (Aim 1a); and using increasingly β1-AR (adrenergic receptor) selective blockers (atenolol and nebivolol), to better define the β-adrenergic receptor selectivity (β1 versus β2) in the regulation of bone turnover by sympathetic outflow in humans.

ELIGIBILITY:
* Inclusion Criteria:

  * at least 5 yrs since their last menses
  * Follicle Stimulating Hormone (FSH) > 20 IU/L
* Exclusion Criteria:

  * Abnormality in any of the screening laboratory studies
  * Presence of significant liver or renal disease
  * Malignancy (including myeloma)
  * Malabsorption
  * Diabetes
  * Hypoparathyroidism
  * Hyperparathyroidism
  * Acromegaly
  * Cushing's syndrome
  * Hypopituitarism
  * Severe chronic obstructive pulmonary disease
  * Undergoing treatment with any medications that affect bone turnover, including the following:
* adrenocorticosteroids (> 3 months at any time or > 10 days within the previous yr)
* anticonvulsant therapy (within the previous year)
* pharmacological doses of thyroid hormone (causing decline of thyroid stimulating hormone below normal)
* calcium supplementation of > 1200 mg/d (within the preceding 3 months)
* bisphosphonates (within the past 3 yrs)
* denosumab
* estrogen (E) therapy within the past year
* treatment with a selective E receptor modulator within the past year
* teriparatide within the past yr
* anti-hypertensive therapy

  * Clinical history of osteoporotic fracture (vertebral, hip, or distal forearm
  * Recent (within the past 6 months) fracture
  * Serum 25-hydroxyvitamin D levels of < 20 ng/ml
  * Resting blood pressure >140/90 mm Hg or those with hypotension (systolic blood pressure <110 mm Hg), heart rate < 60 bpm
  * History of asthma

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2017-10-26 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Ratio of serum bone formation to bone resorption marker | 20 weeks
  Serum bone formation marker (PINP)/serum bone resorption marker (CTX)

CONTACTS AND LOCATIONS:
Overall Officials: Sundeep Khosla, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khosla S, Drake MT, Volkman TL, Thicke BS, Achenbach SJ, Atkinson EJ, Joyner MJ, Rosen CJ, Monroe DG, Farr JN. Sympathetic beta1-adrenergic signaling contributes to regulation of human bone metabolism. J Clin Invest. 2018 Nov 1;128(11):4832-4842. doi: 10.1172/JCI122151. Epub 2018 Oct 2. PMID 30153111